CLINICAL TRIAL: NCT02286713
Title: Promoting Informed Decisions About Lung Cancer Screening: Randomized Trial
Brief Title: PCORI-CER-1306-03385 Informed Decisions About Lung Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014-0628; NCI-2014-02492 (Registry Identifier: NCI CTRP); CER-1306-03385 (Other Grant/Funding Number: Patient Centered Outcome Research Institute)
Record Dates: First submitted 2014-11-03; First posted 2014-11-10 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer; Smoking Cessation; Tobacco Use Cessation
Keywords: Lung Cancer Screening; heavy smokers; state-based smoking cessation quitlines; patient decision aid; low-dose computed tomography; LDCT; standard educational information
MeSH Terms: conditions — Lung Neoplasms; Smoking Cessation; Tobacco Use Cessation | interventions — Videotape Recording; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Decision Aid (Active Comparator): Decision Aid study materials including video mailed to participant with 1-week, 3-month, and 6-month Follow-up Assessments
  Interventions: Behavioral: Patient Decision Aid; Behavioral: Follow-Up Assessments: Questionnaires
- Standard Educational Information (Active Comparator): Study materials including education booklet mailed to participant with 1-week, 3-month, and 6-month Follow-up Assessments
  Interventions: Behavioral: Standard Educational Information; Behavioral: Follow-Up Assessments: Questionnaires

INTERVENTIONS:
Behavioral: Patient Decision Aid — Participants will receive study materials including a video to watch about lung cancer screening
  Other Names: Video; DVD
  Arms: Patient Decision Aid
Behavioral: Standard Educational Information — Participants will receive study materials including a booklet to read about lung cancer screening.
  Other Names: Booklet
  Arms: Standard Educational Information
Behavioral: Follow-Up Assessments: Questionnaires — Follow up questions administered via phone and/or mail at 1-week, 3-month, and 6-month
  Other Names: Survey

SUMMARY:
Educational research study where goal is to test educational materials that help people make informed decisions about lung cancer screening.

DETAILED DESCRIPTION:
This is the second phase of a larger project funded by the Patient-Centered Outcomes Research Institute to help heavy smokers make informed decisions about lung cancer screening with low-dose computed tomography (LDCT). The aim of this phase is to compare outcomes for promoting informed screening decisions about lung cancer screening in a randomized trial of patients who smoke recruited through state-based smoking cessation quitlines, where patients will be randomly assigned to the updated patient decision aid or to standard educational materials on lung cancer screening.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 55 to 77 years of age.
2. Participants must speak English.
3. Current smoker or quit smoking within the past 15 years.
4. At least a 30 pack-year smoking history.

Exclusion Criteria:

1) History of lung cancer.

Ages: 55 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Volk, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- Information and Quality Healthcare (IQH), Ridgeland, Mississippi, United States

REFERENCES:
- [Derived] Volk RJ, Lowenstein LM, Leal VB, Escoto KH, Cantor SB, Munden RF, Rabius VA, Bailey L, Cinciripini PM, Lin H, Housten AJ, Luckett PG, Esparza A, Godoy MC, Bevers TB. Effect of a Patient Decision Aid on Lung Cancer Screening Decision-Making by Persons Who Smoke: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jan 3;3(1):e1920362. doi: 10.1001/jamanetworkopen.2019.20362. PMID 32003822
- [Derived] Lowenstein LM, Escoto KH, Leal VB, Bailey L, Bevers TB, Cantor SB, Cinciripini PM, Jacobs LE, Esparza A, Godoy MC, Housten AJ, Lin H, Luckett P, Munden RF, Rabius V, Volk RJ. Randomized trial of a patient-centered decision aid for promoting informed decisions about lung cancer screening: Implementation of a PCORI study protocol and lessons learned. Contemp Clin Trials. 2018 Sep;72:26-34. doi: 10.1016/j.cct.2018.07.007. Epub 2018 Jul 20. PMID 30010085
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2015 to September 2016 from tobacco quitline new and former callers.
Pre-assignment Details: After consent participants completed baseline assessments prior to randomization.
Period: One Week Follow-Up
Arm/Group | Patient Decision Aid | Standard Educational Information
Started | 259 | 257
Completed | 235 | 233
Not Completed | 24 | 24
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 17 | 21
Not completed — Withdrawal by Subject | 6 | 3
Period: Three Month Follow-Up
Arm/Group | Patient Decision Aid | Standard Educational Information
Started | 252 | 254
Completed | 224 | 228
Not Completed | 28 | 26
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 26 | 24
Not completed — Withdrawal by Subject | 1 | 1
Period: Six Month Follow-Up
Arm/Group | Patient Decision Aid | Standard Educational Information
Started | 250 | 252
Completed | 218 | 225
Not Completed | 32 | 27
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 30 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Decision Aid | Standard Educational Information | Total
Number analyzed (Participants) | 259 | 257 | 516
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 190 | 180 | 370
  >=65 years | 69 | 77 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (5.0) | 61.7 (5.8) | 61.6 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 163 | 320
  Male | 102 | 94 | 196
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Black or African American | 62 | 76 | 138
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Hispanic or Latino | 7 | 1 | 8
  White | 185 | 177 | 362
  Refused | 0 | 1 | 1
  More than one race | 1 | 1 | 2
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 259 | 257 | 516
Participant Pack-Year Smoking History [Median (Inter-Quartile Range); unit: pack-years] — Pack-year smoking history, where one pack-year is equivalent to smoking one pack of cigarettes daily (20 cigarettes) for one year. A 30-pack-year smoking history is an eligibility criterion for lung cancer screening.
  pack-years | 47.0 [40.0 to 63.0] | 49.0 [40.0 to 63.8] | 48.0 [40.0 to 63.0]
Participant Education Level [Count of Participants; unit: Participants]
  Less than High School | 41 | 36 | 77
  Graduated high school/GED | 72 | 77 | 149
  Some college/Trade school | 107 | 105 | 212
  Graduated college or more | 39 | 39 | 78
Participant Health Insurance Status [Count of Participants; unit: Participants]
  Has insurance | 239 | 230 | 469
  Does not have insurance | 20 | 27 | 47

OUTCOME MEASURES:

1. Primary Outcome: Mean Value: Preparation for Decision Making© Scale
Description: The Preparation for Decision Making© Scale assesses a patient's perception of how useful a decision aid or other decision support intervention is in preparing the respondent to communicate with their practitioner at a consultation visit and making a health decision. The scale is scored by summing the 10 items and dividing by 10. Scores are then converted to a 0-100 scale by subtracting 1 and multiplying by 25. Higher scores indicate higher perceived level of preparation for decision making. For this study, researchers used the patient version of the Preparation for Decision Making© scale, adapted for Lung Cancer Screening (LCS) context.
Time Frame: Assessment at 1-week follow-up.
Population: Of participants providing data at the 1-week follow-up, seventeen(17) of the participants did not answer the scale items and were therefore dropped from analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Decision Aid | Standard Educational Information
Number analyzed (Participants) | 227 | 224
units on a scale | 79.4 (17.7) | 69.4 (22.7)

2. Primary Outcome: Mean Value: Informed Subscale of the Decisional Conflict Scale©
Description: A 3-item subscale that measures the degree to which the patient feels informed in making a decision about lung cancer screening. Total scores range from 0 (feels extremely informed) to 100 (feels extremely uninformed) related to making a decision. The scale was adapted for the LCS context.
Time Frame: Assessment at 1-week follow-up.
Population: All participants providing data at the 1-week follow-up where one participant in the Decision Aid Arm did not answer the scale questions and was dropped from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Decision Aid | Standard Educational Information
Number analyzed (Participants) | 234 | 233
units on a scale | 27.1 (25.9) | 42.1 (30.8)

3. Primary Outcome: Mean Value: Values Clarity Subscale of the Decisional Conflict Scale©
Description: A 3-item subscale that measures the degree to which the patient feels clear about his or her values related to the lung cancer screening decision, including values about the harms and benefits. Total scores range from 0 (feels extremely clear about personal value for benefits and risks/side effects of screening) 100 (feels extremely unclear about personal value for benefits and risks/side effects of screening) related to making a decision. The scale was adapted for the LCS context.
Time Frame: Assessment at 1-week follow-up.
Population: Of participants providing data at the 1-week follow-up, one participant in the Standard Educational Information group did not answer the Values Clarity Subscale questions and was dropped from the analysis and where one participant in the Decision Aid Arm did not answer the scale questions and was dropped from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Decision Aid | Standard Educational Information
Number analyzed (Participants) | 234 | 232
units on a scale | 17.6 (26.2) | 31.7 (32.8)

4. Secondary Outcome: Mean Value: Knowledge of Lung Cancer Screening
Description: A 12-item, self-report measure of the patient's knowledge of facts related to lung cancer and lung cancer screening, including the harms and benefits of testing. The knowledge scale yields a single score, representing the percentage of correct responses (ranging from 0% to 100% correct). Higher scores indicate greater knowledge.
Time Frame: One week to 6 months, assessments at 1-week, 3-months and 6-months follow-up.
Population: For the participants providing data at the 1-week follow-up, no data was missing in either group.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Patient Decision Aid | Standard Educational Information
Number analyzed (Participants) | 235 | 233
percentage of correct responses
  One-week | 57.5 (21.8) | 40.1 (17.1)
  3-Months: number analyzed (Participants) | 224 | 228
  3-Months | 44.4 (19.6) | 35.9 (16.9)
  6-Months: number analyzed (Participants) | 218 | 225
  6-Months | 49.9 (17.8) | 40.0 (18.1)

ADVERSE EVENTS:
Time Frame: Adverse event data collected through 6 months participation.
Arm/Group | Patient Decision Aid | Standard Educational Information
All-Cause Mortality (participants affected / at risk) | 4/259 | 1/257
Serious Adverse Events (participants affected / at risk) | 0/259 | 0/257
Other Adverse Events (participants affected / at risk) | 0/259 | 0/257

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT02286713/Prot_SAP_000.pdf